CLINICAL TRIAL: NCT00706342
Title: A Phase II, Open-Label, Efficacy and Safety, Ascending Dose, Pilot Study of be Fostamatinib Disodium/R935788 for the Treatment of Adult Refractory Immune Thrombocytopenic Purpura
Brief Title: Pilot Study of Fostamatinib Disodium/R935788 for the Treatment of Adult Refractory Immune Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4300C00022; C-935788-007 (Other: Rigel Pharmaceuticals)
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
Keywords: Adult Refractory Immune Thrombocytopenic Purpura (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Fostamatinib Disodium / R935788

INTERVENTIONS:
Drug: Fostamatinib Disodium / R935788 — R935788 tablets
  Other Names: R788

SUMMARY:
The purpose of this study is to determine whether Fostamatinib Disodium is safe and effective in the treatment of Adult Refractory Immune Thrombocytopenic Purpura (ITP).

DETAILED DESCRIPTION:
Patients with chronic refractory ITP are eligible for a 6- to 12-week therapeutic trial. After 24 months of treatment, patients who continue to demonstrate a sustained response, in the investigator's judgment, will be offered the opportunity to receive ongoing therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be willing and able to give written informed consent by signing an IRB-approved Informed Consent Form prior to admission to this study.
* Patients may be male or female, between the ages of 18 75. Men, if sexually active, must agree to use at least one medically acceptable form of birth control. Women of childbearing potential must have a negative urine pregnancy test, and agree to use two independent methods of birth control, if sexually active.
* Patients must have a diagnosis of chronic refractory ITP for at least 3 months. Chronic refractory ITP is defined as:

  1. Platelet count < 30,000/mm3 consistently for 3 months (except for transient nonsustained responses to various therapeutic regimens). There must be at least three separate platelet counts (below 30,000/mm3) over this period, with at least one extending back to three months or more prior to patient entry into the study.
  2. The following conditions will have been excluded either by history or appropriate laboratory investigation: HIV infection (see below), lymphoproliferative disorders, myelodysplasia, SLE, drug-induced or alloimmune thrombocytopenia, or dysglobulinemias.
  3. The patient must have tried at least two typical regimens for the treatment of ITP (George et al., Blood, 1996; Practice Guidelines, American Society of Hematology). At least 50% of the enrolled patients will not be known to be refractory to IVIg. Patients may or may not have been treated with IVIg in the past.
* Subjects must test negative for HIV, HBV, and HCV by standard serologic tests within the previous six months.

Exclusion Criteria:

* Patients who have a history or presence of substantial or clinically significant respiratory, gastrointestinal, renal, hepatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, dermatological, or other disorders that, in the Investigator's opinion, could affect the conduct of the study or the absorption, metabolism or excretion of the study drug are excluded. Specifically excluded are lymphoma/chronic lymphocytic leukemia, hepatitis, or HIV associated with ITP.
* Patients who have a history of relevant drug hypersensitivity are excluded.
* Patients who have a history of substance abuse, drug addiction or alcoholism are excluded.
* Patients with the following laboratory abnormalities: a leukocyte count < 2,500/mm3, a neutrophil count of < 1,800/mm3, lymphocyte count < 750/mm3, Hgb < 10 g/L, or transaminase levels (ALT, AST) > 1.5xULN are excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — AstraZeneca
Locations (2):
- United States (2):
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Podolanczuk A, Lazarus AH, Crow AR, Grossbard E, Bussel JB. Of mice and men: an open-label pilot study for treatment of immune thrombocytopenic purpura by an inhibitor of Syk. Blood. 2009 Apr 2;113(14):3154-60. doi: 10.1182/blood-2008-07-166439. Epub 2008 Dec 18. PMID 19096013

RESULTS

PARTICIPANT FLOW:
Groups:
- R788 PO: Tablet containing 75mg BID to 225mg BID R788.
Period: Overall Study
Arm/Group | R788 PO
Started | 18
Completed | 0
Not Completed | 18
Not completed — Adverse Event | 3
Not completed — Not responding to treatment | 2
Not completed — Withdrawn due to failure to respond | 1
Not completed — Death | 1
Not completed — Withdrew from the study on his own. | 1
Not completed — Investigator discretion | 2
Not completed — Non-responder Week 12 | 1
Not completed — Ongoing | 6
Not completed — WIthdrawal of consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | R788 PO
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (15.63)
Age, Continuous [Median (Full Range); unit: years]
  Median (Range) | 65 [30 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Summary of Patients Whose Platelet Count Increased by at Least 20,000/mm3 From Baseline to a Total of 30,000/mm3 or More - Week 2
Time Frame: 2 weeks
Population: Number of participants analyzed refers to the number of patients available at this timepoint for analysis.
Measure: Number; unit: Participants
Arm/Group | R788 PO
Number analyzed (Participants) | 17
Participants | 8

2. Primary Outcome: Summary of Patients Whose Platelet Count Increased by at Least 20,000/mm3 From Baseline to a Total of 30,000/mm3 or More - Week 6
Time Frame: 6 Weeks
Population: Number of participants analyzed refers to the number of patients available at this timepoint for analysis.
Measure: Number; unit: Participants
Arm/Group | R788 PO
Number analyzed (Participants) | 15
Participants | 5

3. Primary Outcome: Summary of Patients Whose Platelet Count Increased by at Least 20,000/mm3 From Baseline to a Total of 30,000/mm3 or More - Week 12
Time Frame: 12 Weeks
Population: Number of participants analyzed refers to the number of patients available at this timepoint for analysis.
Measure: Number; unit: Participants
Arm/Group | R788 PO
Number analyzed (Participants) | 10
Participants | 5

4. Primary Outcome: Summary of Patients Whose Platelet Count Increased by at Least 20,000/mm3 From Baseline to a Total of 30,000/mm3 or More - Week 24
Time Frame: 24 Weeks
Population: Number of participants analyzed refers to the number of patients available at this timepoint for analysis.
Measure: Number; unit: Participants
Arm/Group | R788 PO
Number analyzed (Participants) | 7
Participants | 4

5. Primary Outcome: Summary of Patients Whose Platelet Count Increased by at Least 20,000/mm3 From Baseline to a Total of 30,000/mm3 or More - Month 12
Time Frame: 12 Months
Population: Number of participants analyzed refers to the number of patients available at this timepoint for analysis.
Measure: Number; unit: Participants
Arm/Group | R788 PO
Number analyzed (Participants) | 10
Participants | 5

6. Primary Outcome: Summary of Patients Whose Platelet Count Increased by at Least 20,000/mm3 From Baseline to a Total of 30,000/mm3 or More - Month 24
Time Frame: 24 Months
Population: Number of participants analyzed refers to the number of patients available at this timepoint for analysis.
Measure: Number; unit: Participants
Arm/Group | R788 PO
Number analyzed (Participants) | 7
Participants | 2

ADVERSE EVENTS:
Arm/Group | R788 PO
Serious Adverse Events (participants affected / at risk) | 8/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R788 PO (N=18)
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Mouth hemorrhage (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Anoxic encephalopathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R788 PO (N=18)
Blood glucose increased (Investigations) | 13
Blood pressure increased (Investigations) | 13
Aspartate aminotransferase increased (Investigations) | 11
Blood glucose decreased (Investigations) | 11
Blood alkaline phosphatase increased (Investigations) | 8
Alanine aminotransferase increased (Investigations) | 7
Blood lactate dehydrogenase increased (Investigations) | 6
Blood cholesterol increased (Investigations) | 5
Protein total decreased (Investigations) | 5
BLOOD BILIRUBIN DECREASED (Investigations) | 3
BLOOD BILIRUBIN INCREASED (Investigations) | 3
BLOOD CALCIUM DECREASED (Investigations) | 3
BLOOD POTASSIUM DECREASED (Investigations) | 3
BLOOD UREA INCREASED (Investigations) | 3
HEART RATE INCREASED (Investigations) | 3
ANION GAP INCREASED (Investigations) | 2
BILIRUBIN CONJUGATED (Investigations) | 2
BLOOD CALCIUM INCREASED (Investigations) | 2
BLOOD CHLORIDE DECREASED (Investigations) | 2
BLOOD CREATININE INCREASED (Investigations) | 2
BLOOD MAGNESIUM DECREASED (Investigations) | 2
BLOOD SODIUM DECREASED (Investigations) | 2
GLOBULINS INCREASED (Investigations) | 2
WEIGHT INCREASED (Investigations) | 2
BILIRUBIN CONJUGATED INCREASED (Investigations) | 1
BLOOD ALBUMIN DECREASED (Investigations) | 1
BLOOD BILIRUBIN UNCONJUGATED INCREASED (Investigations) | 1
BLOOD CREATININE DECREASED (Investigations) | 1
BLOOD MAGNESIUM INCREASED (Investigations) | 1
BLOOD PHOSPHORUS DECREASED (Investigations) | 1
BLOOD PHOSPHORUS INCREASED (Investigations) | 1
BLOOD POTASSIUM INCREASED (Investigations) | 1
BLOOD SODIUM INCREASED (Investigations) | 1
BLOOD UREA DECREASED (Investigations) | 1
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 13
PETECHIAE (Skin and subcutaneous tissue disorders) | 12
RASH (Skin and subcutaneous tissue disorders) | 6
BLOOD BLISTER (Skin and subcutaneous tissue disorders) | 4
PRURITUS (Skin and subcutaneous tissue disorders) | 2
SKIN HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 2
URTICARIA (Skin and subcutaneous tissue disorders) | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 1
PURPURA (Skin and subcutaneous tissue disorders) | 1
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 12
NAUSEA (Gastrointestinal disorders) | 7
GINGIVAL BLEEDING (Gastrointestinal disorders) | 5
STOMATITIS (Gastrointestinal disorders) | 5
VOMITING (Gastrointestinal disorders) | 5
HAEMORRHOIDS (Gastrointestinal disorders) | 3
ORAL PAIN (Gastrointestinal disorders) | 3
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 2
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 2
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1
DIVERTICULUM (Gastrointestinal disorders) | 1
DYSPEPSIA (Gastrointestinal disorders) | 1
FAECAL INCONTINENCE (Gastrointestinal disorders) | 1
FAECES DISCOLOURED (Gastrointestinal disorders) | 1
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 1
TONGUE BLISTERING (Gastrointestinal disorders) | 1
TONGUE DISORDER (Gastrointestinal disorders) | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 5
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1
HEADACHE (Nervous system disorders) | 8
DIZZINESS (Nervous system disorders) | 3
SOMNOLENCE (Nervous system disorders) | 3
ANOXIC ENCEPHALOPATHY (Nervous system disorders) | 1
MIGRAINE (Nervous system disorders) | 1
MIGRAINE WITH AURA (Nervous system disorders) | 1
FATIGUE (General disorders) | 7
PYREXIA (General disorders) | 5
OEDEMA PERIPHERAL (General disorders) | 4
PAIN (General disorders) | 3
CHEST PAIN (General disorders) | 2
AXILLARY PAIN (General disorders) | 1
CATHETER SITE INFLAMMATION (General disorders) | 1
FACIAL PAIN (General disorders) | 1
INFLAMMATION (General disorders) | 1
INFLUENZA LIKE ILLNESS (General disorders) | 1
LOCAL SWELLING (General disorders) | 1
MEDICAL DEVICE COMPLICATION (General disorders) | 1
MUCOSAL HAEMORRHAGE (General disorders) | 1
NASOPHARYNGITIS (Infections and infestations) | 5
HERPES ZOSTER (Infections and infestations) | 2
INFLUENZA (Infections and infestations) | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
BREAST ABSCESS (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
OSTEOMYELITIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
SINUSITIS (Infections and infestations) | 1
TOOTH ABSCESS (Infections and infestations) | 1
TOOTH INFECTION (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1
GOUT (Metabolism and nutrition disorders) | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1
HYPERTENSION (Vascular disorders) | 3
HAEMORRHAGE (Vascular disorders) | 2
THROMBOSIS (Vascular disorders) | 2
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
HOT FLUSH (Vascular disorders) | 1
VENOUS INSUFFICIENCY (Vascular disorders) | 1
CONTUSION (Injury, poisoning and procedural complications) | 4
SCRATCH (Injury, poisoning and procedural complications) | 1
PALPITATIONS (Cardiac disorders) | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1
EYE HAEMORRHAGE (Eye disorders) | 2
VISION BLURRED (Eye disorders) | 2
CATARACT (Eye disorders) | 1
DRY EYE (Eye disorders) | 1
EYE PAIN (Eye disorders) | 1
OCULAR HYPERAEMIA (Eye disorders) | 1
EAR PAIN (Ear and labyrinth disorders) | 2
DEAFNESS (Ear and labyrinth disorders) | 1
EAR HAEMORRHAGE (Ear and labyrinth disorders) | 1
HYPOACUSIS (Ear and labyrinth disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 1
PROSTATITIS (Reproductive system and breast disorders) | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1
BREAST PAIN (Reproductive system and breast disorders) | 1
BENIGN GASTROINTESTINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ANXIETY (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
DYSURIA (Renal and urinary disorders) | 1
POLLAKIURIA (Renal and urinary disorders) | 1
URINE ABNORMALITY (Renal and urinary disorders) | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less